CLINICAL TRIAL: NCT03752060
Title: The Clinical Utility of Resistance Training for Improving Cardiovascular Disease Risk in Post-Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ED18101
Record Dates: First submitted 2018-08-15; First posted 2018-11-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Risk Factor; Menopause Related Conditions; Neuromuscular Function; Aerobic Capacity; Inflammation
Keywords: post-menopause; women; post-prandial; metabolic function; cardiovascular function; muscle; body composition; angiogenesis
MeSH Terms: conditions — Inflammation | interventions — Resistance Training; Exercise

STUDY DESIGN:
Intervention Model Description: Following enrollment, participants will complete familiarization and be randomly assigned to an aerobic training (AT; n = 20), a resistance training (RT; n = 20), or a control (CON; n = 20) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Training Group (Experimental): These participants will participate in a progressive resistance training program three times per week on non-consecutive days for 16 weeks. During each session, participants will perform the following exercises: supine bench press, lat pulldown, lateral raise, seated row, leg press, leg extension, leg curl, biceps curl, and triceps extension. The exercises will be completed such that upper body and lower body exercises are alternated throughout each session. During the Weeks 1-4 of training, the subjects will complete two sets of 15 repetitions for each exercise at approximately 50% of their one-repetition maximum (1RM). During Weeks 5-8 of training, the subjects will complete three sets of 12 repetitions at approximately 60% 1RM. During Weeks 9-12, the subjects will complete four sets of 12 repetitions at approximately 60% 1RM. During Weeks 13-16 of training, the subjects will complete 4 sets of 10 repetitions at approximately 70% 1RM.
  Interventions: Behavioral: Resistance Exercise
- Aerobic Training Group (Active Comparator): Women randomized to the AT group will engage in aerobic exercise training that complies with ACSM recommendations10. Specifically, women will complete walking or stationary cycling sessions 5 times per week for 16 weeks. Heart rate data from the pre-intervention VO2peak tests (described below) will be used to estimate each participant's target training heart rate. Like the RT regimen, the AT intervention will be progressive in nature. During the first half of the intervention period, duration will increase by 5 minutes every 2 weeks, from 30 min to 45 min. In the second phase of the intervention, duration will remain constant at 45 min, but intensity will increase from 50% to 65% of heart rate reserve (HRR). Exercise sessions will take place on a treadmill and/or cycle ergometer.
  Interventions: Behavioral: Aerobic Exercise
- Control Group (No Intervention): The control group will complete all baseline and post-testing, but will not complete any training for the 16 weeks between the baseline and post-testing sessions. These participants will also be instructed to maintain their current dietary and physical activity habits (see Lifestyle Controls section). All participants in the control group will also be provided an opportunity to come to the laboratory for two weeks after they have completed the study to receive instruction regarding resistance and/or aerobic training exercise prescription, and to complete supervised resistance and/or aerobic exercise training.

INTERVENTIONS:
Behavioral: Resistance Exercise — Women assigned to the resistance exercise training group will complete progressive, full-body resistance exercise 3 times per week for 16 weeks.
  Arms: Resistance Training Group
Behavioral: Aerobic Exercise — Women assigned to the aerobic exercise training group will complete progressive, aerobic exercise 5 times per week for 16 weeks. The aerobic training will progress first in duration, and then in intensity.
  Arms: Aerobic Training Group

SUMMARY:
Given the heightened cardiovascular disease (CVD) risk in post-menopausal women, studies are needed to explore novel, feasible methods for reducing risk in this population. Based on prior data, primarily in other populations, progressive resistance training is a promising candidate. This project will test the effectiveness of a practical, progressive resistance training regimen for lowering numerous CVD risk factors compared to both aerobic training and no exercise in post-menopausal women.

DETAILED DESCRIPTION:
The number of women living with cardiovascular disease (CVD) is greater than for men and CVD is the leading cause of death for women. Post-menopausal women are a particularly vulnerable population in terms of adverse cardiovascular indicators and outcomes. Specifically, they exhibit greater visceral adipose tissue, fasting and postprandial glucose, total cholesterol (Total-C), fasting insulin, and systolic blood pressure, and are at increased risk for coronary heart disease compared to pre-menopausal women. There is also evidence that cardiovascular indicators (i.e., triglycerides, low high-density lipoprotein cholesterol (HDL-C), etc) are stronger risk predictors in women than men. Despite the staggering rates of CVD in post-menopausal women, as noted by the American Heart Association (AHA), CVD remains understudied in this population. Numerous studies have demonstrated the cardioprotective effects of exercise. However, these studies have largely featured younger individuals, primarily men, undergoing aerobic exercise training. Findings in recent years have indicated the potential benefits of resistance training beyond improving muscular size or strength, such as improved aerobic fitness, central adiposity, glycemic control, and cholesterol profiles. However, large clinical gaps have been noted for women with regard to the effects of resistance training on cardiovascular health. Thus, there is a clear need to assess the cardioprotective effects of progressive exercise training in post-menopausal women.

SPECIFIC AIMS:

1. To test the hypothesis that realistic full-body progressive resistance training improves markers of (a) cardiovascular health and (b) body composition and muscular health in post-menopausal women versus a low physical-activity control.

   A. The primary markers of cardiovascular health to be assessed are aerobic capacity, fasting and postprandial metabolic and inflammatory responses, vascular function via flow-mediated dilation (FMD) and markers of angiogenesis.

   B. The primary body composition and muscle function variables to be assessed are muscle size, isometric and dynamic muscle strength, lean body mass, percent body fat, and abdominal adiposity.
2. To compare the effects of realistic, full-body progressive resistance training in post-menopausal women versus moderate-intensity aerobic exercise, the standard exercise prescription for cardiovascular health, on the cardiovascular, body composition, and muscular health outcomes listed above in 1A. and B.

ELIGIBILITY:
Inclusion Criteria:

* provide written and dated informed consent to participate in the study; (2) be willing and able to comply with the protocol
* be willing and able to comply with the protocol
* be a female between the ages of 45 and 65, inclusive
* be postmenopausal for ≥ 1 year
* be in good health and free from chronic cardiovascular, pulmonary, or musculoskeletal disease as determined by a health history questionnaire
* have a BMI between 18.5 and 40.0, inclusive; and
* answer no to all questions on the PAR-Q for people aged 15 to 69, which are as follows:

  1. Has your doctor ever said that you have a heart condition and that you should only do physical activity recommended by a doctor?
  2. Do you feel pain in your chest when you do physical activity?
  3. In the past month, have you had chest pain when you were not doing physical activity?
  4. Do you lose your balance because of dizziness or do you ever lose consciousness?
  5. Do you have a bone or joint problem that could be made worse by a change in physical activity?
  6. Is your doctor currently prescribing drugs for your blood pressure or heart condition? Do you know of any other reason why you should not do physical activity?

Exclusion Criteria:

* are currently prescribed and/or taking lipid-lowering medications
* are participating in another clinical trial within thirty days prior to enrollment

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic Capacity | A week 0 and immediately after the 16-week intervention period
  Participants will complete a maximal aerobic capacity test to determine VO2peak. The results of this test will be used to determine exercise intensity of the AT training condition, as well as serve as a primary end-point from pre- to post-intervention.
  In brief, participants will start the test at 25 W pedaling between 60-80 rpm, and the workload will be increased by 25 W each minute thereafter. Participants will exercise until they reach volitional fatigue, and can no longer maintain a pedal cadence greater than 60 rpm for 5 consecutive revolutions. Expired gases will be measured throughout the exercise testing via a metabolic cart and heart rate will be assessed using a wireless system.

SECONDARY OUTCOMES:
Change in Metabolic and Inflammatory responses to a Meal Tolerance Test (MTT) | A week 0 and immediately after the 16-week intervention period
  Participants will arrive in the laboratory following a 10 h overnight fast and having abstained from exercise for 48 h. An indwelling 24-gauge safelet catheter (Exel International; Redondo Beach, CA) will be inserted into a forearm vein by a phlebotomist (Dr. Emerson), and a slow infusion (~1 drip/s) of 0.9% NaCl solution will be initiated. A baseline blood draw will be taken to measure fasting metabolic and inflammatory markers. Next, participants will consume a HFM consisting of pie that is 63% fat, 34% carbohydrate, and 3% protein. The amount of pie consumed by each participant is based on body mass (12 kcal/kg). Participants will eat the same HFM pre- and post-intervention. Blood draws will be taken each hour for 6 h post-HFM to characterize the metabolic (TG, glucose, Total-C, HDL-C, LDL-C) and inflammatory and angiogenic (CRP, IL-6, IL-1β, VEGF-A, and VEGF-C) response.
Changes in Vascular Function | A week 0 and immediately after the 16-week intervention period
  Flow-mediated dilation, which will be used to evaluate vascular function, will be assessed via Doppler ultrasound (Linear Array L745 and SonoScape A6 Portable Ultrasound Machine; Shenzhen, China) both fasting and 2 and 4 h post-HFM. After resting in a quiet, dark room for 15 minutes, the brachial artery will be scanned longitudinally slightly above the antecubital crease via a 12 MHz probe. A blood pressure cuff will be inflated to 230-250 mmHg on the proximal portion of the upper arm for 5 minutes, then suddenly released to induce hyperemia. Vascular measurements will be repeated 45-60 seconds after cuff deflation to determine FMD, which decreases following a HFM.
Changes in Body Composition | A week 0 and immediately after the 16-week intervention period
  Height and weight will be measured and body composition assessed pre- and post-intervention using a DEXA scan (Hologic Discovery QDR; Marlborough, MA). Specific outcomes will include percent body fat, lean body mass, and abdominal adiposity.

OTHER OUTCOMES:
Changes in Muscle Strength | A week 0 and immediately after the 16-week intervention period
  Muscle strength will be assessed in two ways: [1] estimated one repetition maximum (1RM) for the dynamic constant external resistance exercises utilized during training, and [2] knee extensor and elbow flexor isometric strength testing.
Changes in Ultrasound-based Assessments of Muscle Size | A week 0 and immediately after the 16-week intervention period
  Ultrasound images of the knee extensors and flexors, elbow extensors and flexors, and plantar flexors will be obtained using a portable brightness mode ultrasound imaging device (GE Logiq S8, USA) and multi-frequency linear-array probe in order to assess muscle size. All ultrasound images will be obtained at the same locations along the muscles of interest at pre- and post-testing and analyzed using Image-J Software (NIH, USA, version 1.47).

CONTACTS AND LOCATIONS:
Locations (1):
- 192 Colvin Recreation Center, Stillwater, Oklahoma, United States